CLINICAL TRIAL: NCT01365078
Title: Effects of Stearidonic Acid on Serum Triacylglycerol Concentrations in Overweight and Obese Subjects
Brief Title: Stearidonic Acid and Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Bioriginal Europe / Asia B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: MEC 11-3-029
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Lipid Metabolism Disorders
Keywords: n-3 polyunsaturated fatty acids; Stearidonic acid; Lipid metabolism; Serum triacylglycerol
MeSH Terms: conditions — Lipid Metabolism Disorders | interventions — stearidonic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Echium oil (SDA-rich oil) (Experimental)
  Interventions: Dietary Supplement: Echium oil (SDA-rich oil)
- High-oleic acid sunflower oil (HOSO) (Placebo Comparator): low in SDA
  Interventions: Dietary Supplement: high-oleic acid sunflower oil (HOSO) (low in SDA)

INTERVENTIONS:
Dietary Supplement: Echium oil (SDA-rich oil) — The echium oil will be provided in sachets containing 5 g of oil, and should be taken for six weeks during the experimental period twice a day, i.e. one sachet at lunch and one sachet at dinner
  Other Names: Oil rich in Stearidonic acid
  Arms: Echium oil (SDA-rich oil)
Dietary Supplement: high-oleic acid sunflower oil (HOSO) (low in SDA) — The HOSO will be provided in sachets containing 5 g of oil, and should be taken for six weeks during the control period twice a day, i.e. one sachet at lunch and one sachet at dinner
  Other Names: Oil low in Stearidonic acid
  Arms: High-oleic acid sunflower oil (HOSO)

SUMMARY:
Evidence exists that EPA (eicosapentaenoic acid or C20:5n-3) supplementation can reduce the risk for coronary heart disease. EPA can be synthesized from α-linolenic acid (ALA or C18:3n-3), but conversion is low. It has been suggested that the rate-limiting step for this conversion is the Δ6-desaturation of ALA into stearidonic acid (SDA or C18:4n-3). Thus, providing oils rich in SDA may increase the endogenous synthesis of EPA. This may subsequently lower serum triacylglycerol concentrations, an effect frequently observed after EPA supplementation, especially in people with increased triacylglycerol levels.

The objective is to study the effects of echium oil, rich in SDA on serum triacylglycerol concentrations in healthy overweight and slightly obese men and women. The minor objective is to study the effects of echium oil on the omega-3 index, which is negatively related to cardiovascular risk and defined as the proportion of EPA and DHA in red blood cells.

DETAILED DESCRIPTION:
Using a randomized, double-blind, placebo controlled crossover design, subjects will receive in random order for six weeks with a washout period of at least 14 days, daily 10 g of echium oil or a high-oleic acid sunflower oil (HOSO) as control.

Thirty-six healthy men and women, aged 18-70 yrs, with a body mass index between 25 and 35 kg/m2 will participate. Subjects with an increased BMI are at increased risk to develop hypertriglyceridemia.

During the experimental period, subjects will receive daily one sachet at lunch and one sachet at dinner each providing 5 g of echium oil. During the control period, subjects will receive daily at the same time points sachets with the same amount of HOSO.

The main study parameter is the change in fasting serum triacylglycerol concentrations. The secondary endpoint is the change in the omega-3 index.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-70 years
* Quetelet-index between 25-35 kg/m2
* mean serum triacylglycerol < 3.0 mmol/L

Exclusion Criteria:

* unstable body weight (weight gain or loss >2 kg in the past 3 months)
* indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus
* use of medication or a diet known to affect serum lipid or glucose metabolism
* active cardiovascular disease like congestive heart failure or recent (<6 months) event (acute myocardial infarction, cerebrovascular accident)
* severe medical conditions that might interfere with the study such as epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel diseases and rheumatoid arthritis
* abuse of drugs
* more than 21 alcohol consumptions per week for men and 14 consumptions for women
* not or difficult to venipuncture as evidenced during the screening visits
* use of an investigational product within the previous 30 days
* not willing to stop the consumption of vitamin supplements, fish oil capsules, fatty fish such as salmon, herring, mackerel and sardine or products rich in plant stanol or sterol esters 3 weeks before the start of the study
* not willing to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study and during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
fasting serum triacylglycerol concentrations | Measured in week 1, 3,5 and 6 of the experimental and the control period

SECONDARY OUTCOMES:
omega-3 index | Measured in week 1, 3, 5 and 6 of the experimental and the control period
  The proportion of EPA and DHA in red blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands